CLINICAL TRIAL: NCT03487809
Title: Evaluate the Therapeutic Effect of Inhaled Corticosteroid in Asthmatic Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Academia Sinica, Taiwan (Other)
Responsible Party: Sponsor
Other Study IDs: 201302019RIND
Record Dates: First submitted 2018-03-19; First posted 2018-04-04 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2022-08

CONDITIONS: Asthma
Keywords: Asthma; Inhaled corticosteroid; pharmacogenomics; Therapeutic effect
MeSH Terms: conditions — Asthma | interventions — Budesonide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, peripheral blood mononuclear cell (PBMC), DNA, RNA
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- NTUH: National Taiwan University Hospital, all participants receive Duasma (budesonide, 200mcg/puff)
  Interventions: Drug: Budesonide/Cisclesonide
- FJUH: Fu Jen University Hospital, all participants receive Duasma (budesonide, 200mcg/puff)
  Interventions: Drug: Budesonide/Cisclesonide
- CGH: Cathay General Hospital, all participants receive Alvesco (Ciclesonide, 160mcg/puff)
  Interventions: Drug: Budesonide/Cisclesonide

INTERVENTIONS:
Drug: Budesonide/Cisclesonide — One arm observation study: Duasma 1 puff bid (Budesonide 200mcg bid) or Alvesco 1 puff qd (Ciclesonide 160mcg qd) for participants aged 11 years and younger, Duasma 2 puffs bid (Budesonide 400mcg bid) or Alvesco 1 puff bid(Ciclesonide 160mcg bid) for participants aged 12 years and older

SUMMARY:
Inhaled corticosteroid (ICS) is considered the first line medication for asthma, however, the therapeutic effect is markedly different even in patients with almost similar clinical manifestations. Our study was designed to explore the clinical and genetic factors that may influence the effectiveness of ICS in asthmatic children.

DETAILED DESCRIPTION:
The three major common classes of asthma controller medications include inhaled corticosteroids (ICS), beta-2-agonists and leukotriene antagonists. Among them, ICS was now suggested as the first-line therapy demonstrated in Global Initiative for Asthma guideline updated in 2017.

The response to asthma medication is markedly different even in patients with almost similar clinical manifestations. Despite the wide availability of therapeutic asthma medications and large studies supporting their efficacy, there is significant inter-personal variability in the response to each of the three major classes of asthma medications with a subgroup of patients that have limited disease control, persistent symptoms and exacerbations even under controller medications use. For example, inter-individual variability in therapeutic effectiveness to ICS in both asthma children and adults is significant, with 22 to 60% of patients being classified as non-responders.

Although many factors can contribute to variation in response to therapy effectiveness, such as higher exhaled nitric oxide, higher total eosinophil counts, higher immunoglobulin E, lower forced expiratory volume at one second (FEV1) predicted. and lower concentration of methacholine needed to produce a 20% fall in FEV1 from baseline (PC20), it is still believed that genetic variability can also play an important role. Hence asthma represents a major burden with respect to mortality, morbidity and National Health Insurance costs, searching for appropriate mediations for asthma control is imperative and investigating the effect of genetic variability on therapy response is an important step to develop personalized prescription.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed by asthma specialists, the age of onset was under 10 years old

Exclusion Criteria:

* Children with cancer, major immunological diseases, such as systemic lupus erythematosus (SLE) or Henoch-Schonlein purpura (HSP), rare hereditary diseases, or under severe infection.
* Children who received ICS or oral steroid in recent 4 weeks

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Asthmatic children with mild to moderate severity, tolerable with inhaled corticosteroid device, can receive blood check.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-10-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
FEV1 | 1 month
  change of forced expiratory volume at one second (FEV1) from baseline

SECONDARY OUTCOMES:
PEF | 1 month
  change of peak expiratory flow (PEF) from baseline
Asthma control test | 1 month
  change of subjective symptoms of asthma
Serum biomarkers | 3 months
  change of ICS response related serum biomarkers (S100 calcium binding protein A12, eosinophil-derived neurotoxin, signal-regulatory protein alpha
  ..)
exhaled nitric oxide (eNO) | 1 month
  change of exhaled nitric oxide
exhaled nitric oxide (eNO) | 3 months
  change of exhaled nitric oxide

CONTACTS AND LOCATIONS:
Overall Officials: Yungling Lee, Professor, Principal Investigator — NTUH
Locations (1):
- NTUH, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
Share with other researchers majored in asthma pharmacogenetic study